CLINICAL TRIAL: NCT01936350
Title: Sildenafil Impact on Ventricular Function in Patients With Heart Failure: Randomized Clinical Trial
Brief Title: Sildenafil Impact on Ventricular Function in Patients With Heart Failure
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospital Ana Nery (Other)
Responsible Party: Principal Investigator, Andre Duraes, PhD, Doctor, Hospital Ana Nery
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 05378712.0.0000.0045
Record Dates: First submitted 2013-09-02; First posted 2013-09-06 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-11

CONDITIONS: Heart Failure
Keywords: Heart failure
MeSH Terms: conditions — Heart Failure | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sildenafil (Experimental): 12 patients will be in this group. They will take a sildenafil 50mg.
  Interventions: Drug: Sildenafil
- Placebo (Placebo Comparator): 12 patients will be in this group, they will take placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil — The intervention in this group is the use of sildenafil 50mg; this group will take placebo and will be evaluated by cardiac magnetic resonance before and after the oral use of the drug.
  Arms: Sildenafil
Drug: Placebo — This group will use placebo; this group will take placebo and will be evaluated by cardiac magnetic resonance before and after the oral use of the placebo pill.
  Other Names: Placebo group
  Arms: Placebo

SUMMARY:
Twenty-four patients with known heart failure will be recruited. They will undergo a cardiac magnetic resonance for ventricular analyses and after this first exam they will be randomized to placebo or Sildenafil. After one hour drug intake they will undergo another cardiac magnetic resonance to evaluate the drug impact on right and left ventricular function.

DETAILED DESCRIPTION:
Twenty-four patients with known heart failure will be recruited. They will undergo a cardiac magnetic resonance for ventricular analyses and after this first exam they will be randomized to placebo or sildenafil. After one hour drug intake they will undergo another cardiac magnetic resonance to evaluate the drug impact on right and left ventricular function.

The first and second exams will be performed by the same staff. All patients will be evaluated by two, three and four chambers view. Left and right ventricle quantification analyses will be performed by Argus software.

ELIGIBILITY:
Inclusion Criteria: Patients with heart failure in stable clinical condition compatible with New York Heart Association functional class I to III. Eligibility criteria is consent to participate in the study after receiving detailed information about procedures, possible clinical benefits, and risks.

Exclusion Criteria: patients with new diagnosed lesions during the procedure, eg pulmonary mass and important claustrophobia, low blood pressure ( systolic blood pressure <90 mmHg or diastolic blood pressure <60 mmHg) nitrate or nebivolol use over the last 48 hours, metallic non MRI compatible implantable devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Improvement on ventricular function | one hour
  Patients will undergo a cardiac magnetic resonance to evaluate ventricular function after one hour of sildenafil or placebo use

CONTACTS AND LOCATIONS:
Overall Officials: Andre M Fernandes, Master, Study Director — Hospital Ana Nery - Federal University of Bahia
Locations (1):
- Hospital Ana Neri - MRI unit, Salvador, Estado de Bahia, Brazil

REFERENCES:
- [Derived] Fernandes AM, Andrade AC, Barroso ND, Borges IC, Carvalho-Andrade D, Rodrigues Junior ES, Guimaraes LC, Duraes AR, Borges SM, Aras Junior R. The immediate effect of sildenafil on right ventricular function in patients with heart failure measured by cardiac magnetic resonance: a randomized control trial. PLoS One. 2015 Mar 20;10(3):e0119623. doi: 10.1371/journal.pone.0119623. eCollection 2015. PMID 25793988
- See also: approved by local Institutional Review Board — http://aplicacao.saude.gov.br/plataformabrasil/visao/pesquisador/gerirPesquisa/gerirPesquisa.jsf